CLINICAL TRIAL: NCT04045522
Title: A Multicenter Prospective Real-world Study on Bisphosphonates Targeting Triple-negative Breast Cancer
Brief Title: Study on Bisphosphonates Targeting Triple-negative Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shengjing Hospital (Other)
Collaborators: Liaoning Cancer Hospital & Institute (Other); The People's Hospital of Liaoning Province (Other)
Responsible Party: Principal Investigator, Caigang Liu, Department director, Shengjing Hospital
Other Study IDs: Shengjing_001
Record Dates: First submitted 2019-07-13; First posted 2019-08-05 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Breast Cancer
Keywords: triple-negative breast cancer; zoledronic acid; real-world study
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Zoledronic Acid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Zoledronic Acid — Based on routine treatment, 4 mg zoledronic acid (Novartis Pharma Stein AG, Switzerland, registration No. H20140218) was intravenously administered, once every 3-4 weeks, for 1-2 years.

SUMMARY:
Triple-negative breast cancer has a poor prognosis and lacks effective adjuvant treatment. A number of preclinical and clinical trials have shown that bisphosphonates have direct or indirect anti-tumor activity, and early use of bisphosphonate adjuvant therapy can prevent cancer recurrence and metastasis including bone metastasis and greatly improve the prognosis of cancer patients. Bisphosphonates have the advantages of low cost, low toxicity, and strong tolerance and can be used as an auxiliary treatment for triple-negative breast cancer. The preliminary study found that bisphosphonates can be chimeric with erlotinib, an epidermal growth factor receptor tyrosine kinase inhibitor, which can synergistically inhibit the in vitro tumor formation of cancer (such as non-small-cell lung cancer and breast cancer) cells and the growth of transplanted tumors. Therefore, the purpose of this multi-center prospective real-world study was to further investigate the effects of bisphosphonate adjuvant therapy on breast cancer.

DETAILED DESCRIPTION:
Triple-negative breast cancer lacks expression of estrogen receptor, progesterone receptor, and proto-oncogene HER2 as shown by immunohistochemical examination. Its incidence accounts for 15-25% of that of all breast cancer types. This type of breast cancer lacks the opportunity of endocrine therapy and anti-human epidermal growth factor receptor 2 (HER2) therapy. The main currently available treatment is still chemotherapy. Some patients may choose anti-angiogenic therapy. The prognosis of triple-negative breast cancer is worse than that of other types of breast cancer due to fewer treatment options. Bisphosphonates used to treat bone metastasis of breast cancer have been shown to have anti-tumor effects and can be used as an adjuvant treatment for triple-negative breast cancer. The preliminary study found that bisphosphonates can be chimeric with erlotinib, an epidermal growth factor receptor tyrosine kinase inhibitor, which can synergistically inhibit the in vitro tumor formation of cancer (such as non-small-cell lung cancer and breast cancer) cells and the growth of transplanted tumors. The persistence of tumor stem cells is reportedly the root cause of malignant biological behavior of triple-negative breast cancer. Bisphosphonates may synergistically inhibit triple-negative breast cancer (stem) cells with existing molecular targeted drugs.

Although randomized controlled trials can provide highest-level clinical evidence, the test conditions should be strictly controlled, resulting in a small sample size and short follow-up time. However, real-world studies can include patients with multiple diseases and treatment strategies can be adjusted according to patient's needs and clinical conditions. In addition, a variety of interventions can be simultaneously used to accurately meet patient's needs, so that the research evidence is more clinically useful. Therefore, the purpose of this multi-center prospective real-world study was to investigate the significance of use of bisphosphonates as an adjuvant therapy against breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* developing breast cancer as confirmed by X-ray examination, and cancer tissue was negative for estrogen receptor, progesterone receptor and HER2
* presence of metastatic axillary lymph nodes
* standardized adjuvant therapy
* age over 55 years

Exclusion Criteria:

* pregnant or lactating women
* those allergic to bisphosphonates
* those who are participating in other trials

Ages: 55 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with triple-negative breast cancer who received treatment in Shengjing Hospital of China Medical University, China.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response time | 5 years
  Pathologic complete response is defined as no residual invasive tumor cells in the breast and axillary lymph nodes

SECONDARY OUTCOMES:
Disease-free survival | 5 years
  It refers to the time from the start of the enrollment to the recurrence of the disease or the death of the patient due to disease progression.
Overall survival | 5 years
  The length of time from either the date of diagnosis or the start of treatment for cancer, that patients diagnosed with the disease are still alive.
Incidence of osteoporosis | 5 years
  Osteoporosis is considered to be present when a patient's bone density or bone mineral content is more than 2.5 standard deviations below the mean value of normal adult bone density.
Incidence of bone-related events | 5 years
  Incidence of bone pain, fracture and other bone related events.
Incidence of other distant organ metastasis-related events | 5 years
  Incidence of metastasis to other distant organs such as the lung, liver, bone marrow, brain and ovary.

CONTACTS AND LOCATIONS:
Overall Officials: Caigang Liu, Principal Investigator — Shengjing Hospital
Locations (3):
- China (3):
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Tumor Hospital & Institute, Shenyang, Liaoning
  - People's Hospital of Liaoning Province, Shenyang, Liaoning

IPD SHARING:
Plan to Share IPD: Undecided